CLINICAL TRIAL: NCT00164827
Title: Phase 3 Study on the Use of Capsule Endoscope for Surveillance and Detection of Peptic Ulcer Rebleeding After Therapeutic Endoscopy
Brief Title: Surveillance of Bleeding Peptic Ulcer Using Wireless Capsule Endoscopy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Other Study IDs: CRE-2002-412-T; CUHK4382/03M
Record Dates: First submitted 2005-09-11; First posted 2005-09-14 (Estimated); Last update posted 2005-09-14 (Estimated); Status verified 2005-09

CONDITIONS: Bleeding Peptic Ulcer
MeSH Terms: conditions — Peptic Ulcer Hemorrhage

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

INTERVENTIONS:
Device: Endoscopic placement of Capsule endoscope adjacent to the peptic ulcer

SUMMARY:
To investigate the adjunctive role of "Capsule Endoscope" in continuous endoscopic monitoring and early detection of recurrent ulcer bleeding after endoscopic therapy in patients presenting with bleeding peptic ulcers

DETAILED DESCRIPTION:
Background

Acute gastrointestinal bleeding is a common medical emergency worldwide. In Hong Kong it accounts for about 5% of all admissions through the Accident and Emergency Department1. The most common cause is bleeding from a peptic ulcer.

Ulcers bleed when an artery at the base of the ulcer is eroded, Bleeding from such an eroded artery may be intermittent, as the artery may be plugged by a thrombus. Dislodgement of the clot results in rebleeding. Rebleeding has long been recognized as one of the worse prognosticators for ulcer bleeding and is associated with a 6-10 fold increase in mortality. Rebleeding is associated with a major bleed manifested by hematemesis and hypotension, indicating that a large size vessel has been eroded. Such vessels, and the clot plugging them, may be visible endoscopically and have been named "stigmata of recent haemorrhage". Such stigmata are associated with a higher risk of rebleeding. High-risk stigmata, such as active bleeding, a protuberant "visible vessel", or an adherent clot, are now used to select patients who are liable to rebleed for endoscopic therapy. In recent years, with advances in endoscopic technology and expertise, therapeutic endoscopy has taken over as the first line therapy for bleeding5. Techniques such as injection therapy, thermal coagulation and clip application have been shown to be highly effective in controlling bleeding7.

Rebleeding after endoscopic therapy

Rebleeding is the most important prognostic factor in patients with ulcer haemorrhage. It carries a 10-fold increase in mortality. Rebleeding can be predicted by hematemesis and shock on admission. Before the era of therapeutic endoscopy traditional dogma recommends early surgery to preempt another catastrophic bleed in these patients. With the advent of effective endoscopic haemostasis the place of early surgery is less clear. Indeed a trial at our center indicates that repeat endoscopic therapy can salvage 75% of rebleeding patients without compromising patient safety10.

Scheduled repeat endoscopy at 24 hour intervals have been used to detect and retreat any remaining stigmata11. Such a policy also subjects many patients to unnecessary endoscopy and treatment but has not been shown to improve outcome. Re-endoscopy at 24-hour intervals misses rebleeding that occurs in the interim, but repeated endoscopy at closer intervals is impractical. Some authors has suggested combining clinical endoscopic data in a scoring system to select patients for repeat endoscopic re-treatment, and demonstrated improved outcome in a small series. Others have used Doppler signals in arteries in the ulcer base to predict failures of endoscopic treatment.

Recognition of rebleeding - Use of wireless endoscopy

Clinical rebleeding is usually defined as vomiting of red blood, hemodynamic instability or drop in the hemoglobin level after initial stabilization. These clinical features appear only after a significant amount of blood has been lost. There is, at present, no reliable method of detecting rebleeding in a timely fashion. If there is a reliable early warning system, analogous to ECG monitoring for arrhythmia in patients who has had a myocardial infarction, we may be able to intervene in time to preempt the harmful effects of further major blood loss in a patient who has already bled from the ulcer.

Endoscopy using a pill sized (11mm x 26mm, weight ~ 4 grams) capsule endoscope was first reported by Iddan. The capsule can be swallowed and transmit images from various part of the gastrointestinal tract as the capsule traverses the gastrointestinal tract. The main indication at present is the visualization of the small intestine, especially for locating sources of bleeding that are beyond the range of gastroscopy and colonoscopy. The battery of the capsule lasts for up to 8 hours.

We aimed to use the capsule endoscope to monitor the bleeding peptic ulcer after therapeutic endoscopy in order to detect rebleeding before clinical manifestation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with bleeding peptic ulcers; ulcer actively bleeding or with major stigmata of visible vessels ( protuberant discolorations in ulcer bases) and clots (Forrest I, IIa and IIb ulcers) seen at endoscopy performed within 24 hours of their admissions.
* Endoscopic hemostasis achieved (with defined endpoints).
* Age > 18
* Provision of an informed written consent signed by the patient.

Exclusion Criteria:

* The present of an intercurrent ulcer complication precluding endoscopic treatment such as gastric outlet obstruction or ulcer perforation mandating surgical intervention.
* Patients with clinical suspicion of intestinal obstruction, stricture and fistula.
* Patient with cardiac pacemaker, or any implanted electromedical device.
* Age <18
* Pregnancy
* moribund patients e.g. patients with terminal malignancy
* Patient unable to give written consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2003-01

CONTACTS AND LOCATIONS:
Overall Officials: Enders KW Ng, MD, Principal Investigator — Department of Surgery, Prince of Wales Hospital, The Chinese University of Hong Kong
Locations (1):
- Endoscopy Center, Prince of Wales Hospital, Hong Kong, China